CLINICAL TRIAL: NCT03936868
Title: Tendon Transfer Surgery for Irreversible Radial Nerve Palsy, Does it Help When Expert is Available? Retrospective Cohort From Level-1 Trauma Center in a Metropolitan City.
Brief Title: Tendon Transfer for Irreversible Radial Nerve Palsy, Does it Help?Retrospective Cohort From Level-1 Trauma Center.
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Obada Hasan, FCPS, MRCS, Senior Resident, Aga Khan University
Other Study IDs: 2019-0845-3203
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Radial Palsy
MeSH Terms: conditions — Radial Neuropathy | interventions — Tendon Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tendon transfer for irreversible radial nerve palsy patient: Tendon transfer for irreversible radial nerve palsy patient who had irreversible damage to radial nerve due to trauma with different mechanism especially gun shot injury
  Interventions: Procedure: Tendon transfer

INTERVENTIONS:
Procedure: Tendon transfer — flexor carpi radialis transfer in most of patients and boye-transfer in very few

SUMMARY:
Radial nerve palsy is associated with serious disability jeopardizing the grasp and power grip accountable to the loss of thumb and fingers extension and loss of active wrist extension respectively. There are three aims in the treatment of radial nerve palsy which comprise the restoration of thumb extension and abduction, finger extension and restoration of wrist extension. In this study we measured the functional outcome after tendon transfer for radial nerve palsy aimed to restore the wrist extension, finger extension and thumb extension/abduction. Investigators' objective was to assess the functional outcome after tendon transfer surgery for radial nerve palsy.

DETAILED DESCRIPTION:
Radial nerve palsy is associated with serious disability jeopardizing the grasp and power grip accountable to the loss of thumb and fingers extension and loss of active wrist extension respectively. There are three aims in the treatment of radial nerve palsy which comprise the restoration of thumb extension and abduction, finger extension and restoration of wrist extension. In this study we measured the functional outcome after tendon transfer for radial nerve palsy aimed to restore the wrist extension, finger extension and thumb extension/abduction. Investigators' objective was to assess the functional outcome after tendon transfer surgery for radial nerve palsy. So investigators conducted a retrospective study at Aga Khan University Hospital Karachi comprising records of patients operated for irreversible high radial nerve palsy. Investigators concluded that tendon transfer surgery for radial nerve palsy provides excellent results to restore the lost function and therefore must be considered for patients with no signs of recovery after the nerve repair.

ELIGIBILITY:
Inclusion Criteria:

* All participants including paediatric and adult age group with irreversible radial nerve palsy and patients with radial nerve palsy with time interval of more than 9 months were included.

Exclusion Criteria:

* All participants who underwent radial nerve repair or nerve grafting with or without internal splinting, patients with vascular injuries, muscular dystrophies, CVA (Cerebero-Vascular Accident), Dementia and those with limited followup of less than 3 months were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: participants with presenting due to late consequence of trauma affecting their hand and wrist function due to irreversible damage to radial nerve
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Functional outcome - Range of Motion | 6 months
  Range of Motion at hand and wrist joints, fingers extension, wrist extension

IPD SHARING:
Plan to Share IPD: No
Not having permission from institute.